CLINICAL TRIAL: NCT02903719
Title: The Effect of Phrenic Nerve Block on Postoperative Shoulder Pain in Patients for Liver Resection - a Double Blinded Randomised Controlled Trial.
Brief Title: The Effect of Phrenic Nerve Block on Postoperative Shoulder Pain in Patients for Liver Resection.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eske Kvanner Aasvang (Other)
Responsible Party: Sponsor-Investigator, Eske Kvanner Aasvang, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13001
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Shoulder Pain; Surgery; Nerve Block
Keywords: Phrenic; Nerve block; Postoperative shoulder pain; Liver resection
MeSH Terms: conditions — Shoulder Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): 1. st intervention: A single ultrasound guided perineural injection of Ropivacaine 7,5 mg/ml, 3 ml
  2. nd intervention (approx. 15 minutes after 1st intervention): A single ultrasound guided perineural injection of isotonic saline solution 9 mg/ml, 3 ml
  Interventions: Drug: Ropivacaine
- Group B (Other): 1. st Intervention: A single ultrasound guided perineural injection of isotonic saline solution 9 mg/ml, 3 ml
  2. nd Intervention (approx. 15 minutes after 1st intervention):A single ultrasound guided perineural injection of Ropivacaine 7,5 mg/ml, 3 ml
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — All included patients with a right sided shoulder pain score on a numeric rating scale (NRS) equal to or above 6 and without postoperative exclusion criteria will have two (1st and 2nd intervention) ultrasound guided phrenic nerve blocks performed.
  Other Names: Naropin

SUMMARY:
The aim of this study is to explore whether the use of ultrasound guided phrenic nerve block can reduce the postoperative pain in the shoulder after liver resection. The intervention is directed postoperative to the patients experiencing novel right sided shoulder pain.

DETAILED DESCRIPTION:
Background:

Patients undergoing both laparoscopic and open hepatic surgery often experience shoulder pain in the postoperative period, mostly on the right side.

The mechanism behind referral of pain from surgical sites to the ipsilateral (same side) shoulder is not fully understood. It has been stated, that the sharing of cervical sensory roots, leads the brain to an interpretation that the pain as originating from the ipsilateral shoulder, when the phrenic nerve is stimulated.

The phrenic nerve provides both sensory and motor nerves to the diaphragm, and sensory fibers to parts of the pleura and peritoneum. Furthermore, one anatomical study indicate, that the phrenic nerve on the right side supply the liver capsule with thin sensory nerves. This could also, in part, explain the shoulder pain after liver surgery.

Studies assessing the effect of phrenic block on shoulder pain by surgically applied intrathoracic block of the phrenic nerve, have found a pain reduction, without significant side effects. There are no available studies on the effect of phrenic nerve block after hepatic surgery. Blocking the nerve intraoperatively, as described in thoracic surgery, is not possible during these operations.

Pilot study of the incidence: A recent survey at Rigshospitalet, Denmark, revealed, that 19 out of 60 patients undergoing various types of hepatic surgery, experienced moderate to severe right sided shoulder pain in the post operative care unit. The only semi-effective treatment, has been opioids (morphine), often leading to significant side effects (nausea, vomiting , dizziness) with a potential for an increase in postoperative morbidity. Furthermore, referred shoulder pain affects the respiratory capacity postoperatively.

The investigators have developed a method for applying ultrasound-guided block at the lateral side of the neck, directly at the phrenic nerve where it crosses over the scaleni anterior muscle. The block is done with low volume of local anesthetic (only 3 ml very close to the nerve) aiming to avoid affection of the brachial plexus.

The phrenic nerve block have been performed at right sided shoulder pain in the postoperative care unit with marked effect within a few minutes (small nerve with little perineural insulation).

Trial endpoints:

The idea of the study is to perform a precise, low volume, ultrasound guided nerve block in the patients who experience a severe right sided shoulder pain (NRS >5 on a 0-10 scale) after liver surgery and evaluate the effect of active substance vs. placebo

Furthermore the investigators wish to stablish an evaluation of the duration of the phrenic nerve block when it comes to pain intensity, incidence of referred shoulder pain after liver surgery, and need for opioid and to evaluate the effect of the block on the lung function.

The study results will be described in a primary publication regarding the primary outcome, and a secondary publication regarding the incidence of acute respiratory and ventilatory affection observed in the PACU in patients undergoing open liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18.
* Patients scheduled for liver resection.
* Ability to give informed consent.

Exclusion Criteria:

* Participation in another clinical trial, dealing with pain or management of pain, which could affect this trial, evaluated by the investigator.
* Inability to talk and understand danish
* Drug or alcohol abuse
* Pregnancy
* Congestive heart failure (NYHA class III-IV), or other serious heart disease.
* Chronic obstructive lung disease, moderate or severe degree, or other significant lung disease
* Chronic or acute shoulder pain prior to surgery.
* Body Mass Index above 35.
* Infection at the site of the injection
* Allergy to ropivacaine

Postoperative:

* Shoulder pain score < 6 assessed on the numeric rating scale (0-10), 15 minutes after arrival in postanaesthetic care unit (PA CU).
* Insufficient epidural analgesia, or lack of epidural analgesia.
* Inability to visualize nervus phrenicus with sonography.
* Cerebral confusion, postoperative delirium or other medical condition hindering study intervention.
* Presence of an investigator with intervention competence is not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Pain measurements on a NRS (Numeric Rating Scale) | 1 hour
  Patients are asked to rate the intensity of their shoulder pain (if any) according to NRS (Numeric Rating Scale) from 0-10 (0=no pain, 10=the worst pain imaginable). For patients receiving the intervention they are asked to rate the intensity of their pain 15 minutes after the 1st intervention.

SECONDARY OUTCOMES:
Lung function assessed by Spirometry | 1 day
  Lung function evaluated with spirometry (FEV1, FVC og VC) just prior to
  1st intervention (baseline), compared to lung function after 1st intervention or 2nd intervention. Patients receiving the interventions get their lung function measured 3 times after the interventions. Patients excluded postoperatively get their lung function measured once.
Lung function assessed by arterial blood gas | 1 hour
  Lung function evaluated with arterial blood gas (paO2, paCO2) just prior to 1st intervention (baseline), compared to lung function after 1st intervention or 2nd intervention. Lung function is also evaluated with arterial blood gas one hour after 2nd intervention.
Duration of surgery compared to shoulder pain | 1 hour
  Duration of surgery compared to shoulder pain just prior to 1st intervention. The intensity of pain is measured according to NRS (0-10, 0=no pain, 10=worst pain imaginable).
Number of included patients with low pain score (NRS) after interventions. | 1 hour and 15 minutes
  Number of included patients with a pain score (NRS) between 0 and 3 after 1st intervention or 2nd intervention.
Number of patients with respiratory affection | 1 day
  Number of included patients with respiratory affection, if defined as this in the medical chart.
Number os patients treated with opioid | 2 hours
  Number of included patients treated with opioid and the amount of used opioid in morphine equivalence.
Prevalence of respiratory and cardiovascular events amon included and excluded patients. | 30 days
  Prevalence of respiratory og cardiovascular events until discharge when defined as this in medical chart and prevalence of readmission obtained from the Danish National Hospital Registry.
Pain measurements 24 hours after the 1st intervention. | 24 hours
  Patients are asked to rate the intensity of their shoulder pain according to NRS (numeric rating scale 0-10) 24 hours after the 1st intervention.
Pain measurements on a NRS (Numeric Rating Scale) | 2 hours
  Patients are asked to rate the intensity of their shoulder pain (if any) according to NRS (Numeric rating scale) from 0-10 (0=no pain, 10=the worst pain imaginable). For patients receiving the intervention they are asked to rate the intensity of their pain +2, +5, +10 and +60 minutes after the 1st intervention and +2, +5, +10 and +15 after the 2nd intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided